CLINICAL TRIAL: NCT04321889
Title: Randomized Double-blind Controlled Trial to Evaluate the Efficacy of Defurocumarinized Bergamot Loaded in a Nanotechnological System for the Release of Essential Oil in the Treatment of Agitation in Severe Dementia Patients.
Brief Title: Efficacy of Defurocumarinized Bergamot in the Treatment of Agitation in Severe Dementia Patients.
Acronym: BEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: S.Anna Rehabilitation Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISA-BEO092019
Record Dates: First submitted 2020-03-10; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Severe Dementia; Stroke
MeSH Terms: conditions — Dementia; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo clinical trial for parallel groups to evaluate the clinical efficacy of defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of a cream in the treatment of agitation, in patients of both sexes with severe dementia diagnosis. Subjects will be eligible if they meet all inclusion criteria. A total of 134 patients will be enrolled, randomized, in a 1:1 ratio, to treatment with defurocumarinized bergamot loaded in a nanotechnological release system or placebo.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEO (Experimental): Subjects of both sexes of age >65 years who have received diagnosis of severe dementia and clinically relevant agitation hospitalized in the enrolment center.
  Interventions: Device: defurocumarinized bergamot loaded in a nanotechnological essential oil release system
- Placebo (Placebo Comparator): Subjects of both sexes of age >65 years who have received diagnosis of severe dementia and clinically relevant agitation hospitalized in the enrolment center.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: defurocumarinized bergamot loaded in a nanotechnological essential oil release system — Patients will be treated either with placebo cream or with defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of cream 2 times a day for 4 weeks. The subject will be monitored throughout the treatment and for at least 4 weeks after the end of the treatment.
  Arms: BEO
Other: Placebo — nanotechnological system loaded with placebo cream
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of defurocumarinized bergamot in the treatment of agitation in severe dementia patients. Bergamot essential oil (BEO), able to modulate the endogenous, peripheral and central opioid system involved in painful states, has developed in models of inflammatory pain and neuropathic pain; it is also effective when administered by inhalation.

Participants in the study will be divided into 2 parallel groups, one treatment group and one placebo, to evaluate the clinical efficacy of defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of a cream in the treatment of agitation, in in Over-sixty-five-year-old patients of both sexes diagnosed with severe dementia.

DETAILED DESCRIPTION:
According to the World Alzheimer's Report 2018, 50 million people worldwide suffer from dementia and it is estimated that this number will triple by 2050.

Very often people with dementia suffer from comorbidities accompanied by chronic, inflammatory and neuropathic pain, often under-diagnosed through psychological and behavioral symptoms of dementia such as agitation and aggression. The therapy of neuropsychiatric symptoms of dementia is currently based on the use of atypical antipsychotics that are actually present in the short term and may induce important side effects.

This study evaluates the efficacy of defurocumarinized bergamot in the treatment of agitation in severe dementia patients. Bergamot essential oil (BEO), able to modulate the endogenous, peripheral and central opioid system involved in painful states, has developed in models of inflammatory pain and neuropathic pain; it is also effective when administered by inhalation. To solve this problem, this clinical trial will use defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of an odourless cream indistinguishable from placebo cream.

Participants in the study will be divided into 2 parallel groups, one treatment group and one placebo, to evaluate the clinical efficacy of defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of a cream in the treatment of agitation, in in Over-sixty-five-year-old patients of both sexes diagnosed with severe dementia.

The rationale of this clinical trial is based on three fundamental points:

1. Preclinical research has proven, beyond any doubt, a powerful analgesic activity of BEO on inflammatory and neuropathic pain;
2. at present the essential oils needed in aromatherapy for agitation management do not show strong analgesic activity, documented by extensive preclinical evidence;
3. clinical trials that have assessed the efficacy of aromatherapy in neuropsychiatric symptoms associated with dementia suffer from the severe lack of a double-blind according to the most rigorous criteria of clinical trial evaluation. To solve this problem, this clinical trial will use defurocumarinized bergamot loaded in a nanotechnological system of essential oil release in the pharmaceutical form of an odourless cream indistinguishable from placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe dementia by MMSE score<12;
* Signature of informed consent by a family member/caregiver/support administrator;
* The use of authorised and concomitant therapies for the treatment of agitation is permitted.

Exclusion Criteria:

-Positive remote case history for pre-existing neurological or psychiatric disabling conditions

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment of agitation | up to 6 weeks after the end of treatment
  To evaluate the clinical efficacy of defurocumarinized bergamot l in the treatment of agitation in patients with severe dementia by determination of the Cohen-Mansfield Agitation Inventory (CMAI)score. CMAI is a 29-item scale widely used to assess agitation.

SECONDARY OUTCOMES:
Duration of the effect on agitation | 6 weeks after the end of treatment
  Carry out a follow-up following suspension of the treatment with defurocumarinized bergamot loaded in a nanotechnology essential oil release system to assess the duration of the effect on agitation, using Cohen-Mansfield Agitation Inventory (CMAI) score. CMAI is a 29-item scale widely used to assess agitation.
clinical efficacy on pain | 6 weeks after the end of treatment
  Determine the clinical efficacy of defurocumarinized bergamot, loaded in a nanotechnological system of essential oil release in the pharmaceutical form of a cream, on pain in patients with severe dementia by determining the weekly score of the Mobilization-Observation-Behaviour-Intensity-Dementia (MOBID)-2 pain assessment scale. MOBID-2 is an extended version of the MOBID pain scale and consists of two parts: Part 1 is the previous MOBID and is used for the assessment of musculoskeletal pain through the observation of painful behaviour when performing five guided movements of different parts of the body in order to assign a score to the pain intensity; Part 2 is used for the assessment of pain from internal organs, head and skin, through behavioural indicators of pain and pain localization on the pain site illustrations.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Tonin, MD, Principal Investigator — S.Anna Rehabilitation Insitute

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual partecipant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the end of the study
Access Criteria: Data access request will be reviewed by an internal audit committee in conjunction with a panel of university experts

REFERENCES:
- [Background] Scuteri D, Rombola L, Morrone LA, Bagetta G, Sakurada S, Sakurada T, Tonin P, Corasaniti MT. Neuropharmacology of the Neuropsychiatric Symptoms of Dementia and Role of Pain: Essential Oil of Bergamot as a Novel Therapeutic Approach. Int J Mol Sci. 2019 Jul 6;20(13):3327. doi: 10.3390/ijms20133327. PMID 31284573
- [Background] Scuteri D, Morrone LA, Rombola L, Avato PR, Bilia AR, Corasaniti MT, Sakurada S, Sakurada T, Bagetta G. Aromatherapy and Aromatic Plants for the Treatment of Behavioural and Psychological Symptoms of Dementia in Patients with Alzheimer's Disease: Clinical Evidence and Possible Mechanisms. Evid Based Complement Alternat Med. 2017;2017:9416305. doi: 10.1155/2017/9416305. Epub 2017 Mar 30. PMID 28465709
- [Background] Scuteri D, Crudo M, Rombola L, Watanabe C, Mizoguchi H, Sakurada S, Sakurada T, Greco R, Corasaniti MT, Morrone LA, Bagetta G. Antinociceptive effect of inhalation of the essential oil of bergamot in mice. Fitoterapia. 2018 Sep;129:20-24. doi: 10.1016/j.fitote.2018.06.007. Epub 2018 Jun 12. PMID 29906556
- [Background] Sakurada T, Mizoguchi H, Kuwahata H, Katsuyama S, Komatsu T, Morrone LA, Corasaniti MT, Bagetta G, Sakurada S. Intraplantar injection of bergamot essential oil induces peripheral antinociception mediated by opioid mechanism. Pharmacol Biochem Behav. 2011 Jan;97(3):436-43. doi: 10.1016/j.pbb.2010.09.020. Epub 2010 Oct 13. PMID 20932858
- [Background] Sakurada T, Kuwahata H, Katsuyama S, Komatsu T, Morrone LA, Corasaniti MT, Bagetta G, Sakurada S. Intraplantar injection of bergamot essential oil into the mouse hindpaw: effects on capsaicin-induced nociceptive behaviors. Int Rev Neurobiol. 2009;85:237-48. doi: 10.1016/S0074-7742(09)85018-6. PMID 19607974
- [Background] Berliocchi L, Russo R, Maiaru M, Levato A, Bagetta G, Corasaniti MT. Autophagy impairment in a mouse model of neuropathic pain. Mol Pain. 2011 Oct 24;7:83. doi: 10.1186/1744-8069-7-83. PMID 22023914
- [Derived] Scuteri D, Pagliaro M, Mantia I, Contrada M, Pignolo L, Tonin P, Nicotera P, Bagetta G, Corasaniti MT; Pilot BRAINAID Trial investigators. Efficacy of therapeutic intervention with NanoBEO to manage agitation and pain in patients suffering from severe dementia: a pilot clinical trial. Front Pharmacol. 2024 Aug 1;15:1417851. doi: 10.3389/fphar.2024.1417851. eCollection 2024. PMID 39148533
- [Derived] Scuteri D, Sakurada S, Sakurada T, Tonin P, Bagetta G, Nicotera P, Corasaniti MT. Requirements for Translation in Clinical Trials of Aromatherapy: The Case of the Essential Oil of Bergamot (BEO) for Management of Agitation in Severe Dementia. Curr Pharm Des. 2022;28(20):1607-1610. doi: 10.2174/1381612828666220509152029. PMID 35579159